CLINICAL TRIAL: NCT00576615
Title: CNS Targets of Propofol's Hypnotic and Memory Effects
Brief Title: Propofol's Hypnotic and Memory Effects
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 01-139
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: healthy volunteers; amnesic effects
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: placebo: placebo solution
  Interventions: Drug: Placebo solution
- 2: propofol: propofol
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: Placebo solution — On the day of the study infusion into the vein of a solution containing no drug, Complete about half a dozen memory tasks over the period of the study, each about 5-10 minutes in length, that involve identification of a list of words, or listen to a list of words/tones before, during, and/or after drug infusion. Allow the recording of your brain waves - the faint electrical activity constantly occurring in your brain- using the electroencephalogram (EEG) while completing memory tasks. Allow the imaging of your brain using functional magnetic resonance imaging (MRI), which measures images of water in your brain in a strong magnetic field, while completing memory tasks.
  Groups: 1: placebo
Drug: propofol — On the study day you will receive study drug propofol. Complete about half a dozen memory tasks over the period of the study, each about 5-10 minutes in length, that involve identification of a list of words, or listen to a list of words/tones before, during, and/or after drug infusion.
  Allow the recording of your brain waves - the faint electrical activity constantly occurring in your brain- using the electroencephalogram (EEG) while completing memory tasks. Allow the imaging of your brain using functional magnetic resonance imaging (MRI), which measures images of water in your brain in a strong magnetic field, while completing memory tasks.
  Groups: 2: propofol

SUMMARY:
The purpose of this study is to relate changes in the blood flow in your brain which are measured using magnetic resonance imaging (MRI) to temporary changes in your memory and level of sleepiness while receiving the drug propofol, which is commonly used to induce relaxation or sleepiness for minor surgical procedures. This study will help provide us information which will be useful in understanding which parts of the brain are influenced by these drugs to affect memory and sleepiness.

DETAILED DESCRIPTION:
We wish to seek evidence of a neuroanatomical basis for the separation of the sedative/hypnotic and amnesic effects of propofol by imaging electrophysiologic and regional cerebral blood flow (rCBF) changes to identify these. Our main hypothesis is that there are differing neuroanatomical regions mediating drug-induced sedation and amnesia, and that these can be identified by specific changes in electrophysiology and rCBF. Electrophysiologic changes will be mapped using a validated electroencephalographic (EEG) mapping technique, Low Resolution brain Electromagnetic Tomography (LORETA). (1) Changes in brain activity will be identified with high spatial resolution using magnetic resonance imaging (MRI) and statistical parametric mapping (SPM). (2) To identify key regions out of possibly many exhibiting changes in brain activity during propofol administration, we plan to manipulate drug-induced sedation by using thiopental, a sedative drug with few memory effects active at the same receptors as propofol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal volunteers who show no evidence of neurologic deficit on questionnaire and physical examination
* Females of child-bearing age must be non-pregnant as demonstrated using a pregnancy test, non-lactating, and must be using adequate contraception or be surgically sterile
* Age 18 years to 45 years
* Right hand dominant
* High school education or above(to ensure consistent performance on the memory tests being administered)
* English as native language or equivalent degree of fluency

Exclusion Criteria:

* Any evidence of neurologic deficit including seizures, history of severe head trauma or any previously or current abnormal study of CNS - (eg. MRI, EEG, etc.)
* Any deficit in auditory or visual ability that would prevent performance of the study tasks
* History of claustrophobia
* Any history of hypertension (resting BP >150 systolic, >100 diastolic) or taking anti- hypertensive medication
* Any history of cardiovascular disease including previous myocardial infarction, arrhythmia, heart valve disease, or cardiac murmur
* Significant pulmonary, renal, gastrointestinal, or endocrine metabolic disease which in the opinion of the investigator would complicate the goals of this study
* Allergy to propofol, thiopental, eggs or history of acute intermittent porphyria, history of severe allergic reaction (e.g. anaphylactic shock)
* History of substance abuse
* Currently taking centrally acting medications (benzodiazepines or other anxiolytics, antidepressants, antipsychotic agents, or agents affecting the cerebral vasculature)
* Any one who is not NPO for at least 6 hours
* Any implant incompatible with MR scanning
* Anyone who, in the opinion of the investigators, would be unwilling or unable to tolerate the procedures and/or comply with the task instructions
* Body Mass Index (BMI) > 30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: MSKCC clinics
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2002-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate the persistence of defined stimulation-related changes in brain activity during various levels of propofol and thiopental sedation. | fifteen hours over several different days

SECONDARY OUTCOMES:
Identify the neuroanatomical regions mediating propofol-induced amnesia and sedation. | fifteen hours over several different days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Veselis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org